CLINICAL TRIAL: NCT00433238
Title: Screening for Mental Health Concerns for at-Risk Community Living Chinese Seniors - a Feasibility Study
Brief Title: Screening for Mental Health Concerns for at-Risk Community Living Chinese Seniors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: WCMSH
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Major Depressive Disorder; Dementia
Keywords: elderly; Chinese; community living; measurement; depression; dementia; Geriatric Depression Scale; MiniCog
MeSH Terms: conditions — Depressive Disorder, Major; Dementia; Depression

INTERVENTIONS:
Behavioral: Participants will be screened for depression and cognitive impairment, then receive screening results.

SUMMARY:
The study is designed to answer the following research questions:

1. Evaluate the acceptability of mental health screening and of the instruments used in a sample of community living Chinese seniors;
2. Determine rates of mental health service utilization in individuals identified at screening as having psychological disturbance;
3. Determine if identifying mental illness and informing participants of screening results and with treatment alternatives alters help-seeking pathways.

The study hypotheses are:

1. This community sample of Chinese seniors will show a higher prevalence of psychological disturbance than their counterparts in the general population;
2. Emotional well-being will be positively correlated with individuals' physical health and social support network.

DETAILED DESCRIPTION:
A convenience sample will be drawn from 6 Congregate Dining (CD) groups in the Chinese community. There are six groups of CD programs run by Yee Hong Centre for Geriatric Care run at different locations in the Greater Toronto Area. The screening will be offered on site at regular CD meetings to participants who have given informed, written consent. All participants will attend a private post-screening interview. Those who score above the threshold for depression and/or cognitive impairment, and who have not previously been diagnosed or treated for these conditions, will be randomly assigned to one of two groups: an intervention group and a usual care group. Participants in the intervention group will receive their screening results at the post-screening interviews and will also be provided with suggestions for possible follow-up. They will be given the option of receiving further psychiatric assessment at the Wellness Centre, or seeking care with their family physician and assisted to obtain further care, if desired. Participants in the intervention group will attend an appointment 3 months after receiving screening results and follow-up options during which the rate of help seeking, rate of confirmed psychiatric diagnoses and types of intervention received will be determined. Participants in the usual care group will not be given screening results at the post-screening interview but will instead attend an appointment 3 months post screening to receive their results and information about follow-up options.

The results of this research will: demonstrate whether community living Chinese elders are at greater risk of psychiatric disorders and demonstrate the need for screening in older Chinese adults living in the community; aid in the development of systematic and targeted community-based screening and outreach to at-risk members of the target population; and help determine if identification of mental health issues and education about treatment resources has any effect on help-seeking for those conditions.

ELIGIBILITY:
Inclusion Criteria:

* capable of providing informed consent
* informed consent

Exclusion Criteria:

* Individuals who are unable to fully understand the nature of the study, its possible risks and benefits and the consequences of providing or withholding consent, and who are, therefore, not capable of providing informed consent will be excluded from the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2007-03

PRIMARY OUTCOMES:
Rate of help seeking in intervention group
Rate of confirmed psychiatric diagnoses in intervention group
Type of intervention received

CONTACTS AND LOCATIONS:
Overall Officials: Joel Sadavoy, M.D., Principal Investigator — Mt. Sinai Hospital, Toronto, Canada
Locations (1):
- Wellness Centre, Toronto, Ontario, Canada